CLINICAL TRIAL: NCT06476665
Title: BESPONSA INJECTION 1MG SPECIAL INVESTIGATION (PEDIATRIC INVESTIGATION)
Brief Title: A Study to Learn About the Safety of BESPONSA Injection in Pediatric Patients With Acute Lymphocytic Leukemia.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1931035; NCT06476665 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about the safety of BESPONSA for pediatric patients. .

BESPONSA is approved for treatment of relapsed or refractory CD22-positive acute lymphocytic leukemia for pediatric patients. A type of leukemia (blood cancer) that comes on quickly and is fast growing. In acute lymphocytic leukemia, there are too many lymphoblasts (early-stage white blood cells) in the blood and bone marrow. Also called ALL.

The registration criteria for this study are:

* Never used BESPONSA before
* <18 years at the start of treatment with BESPONSA

All patients in this study will receive BESPONSA according to the prescriptions.

Patients will be followed up as follow.

* Treatment phase: From the day of treatment initiation (Day 1) to Day 28 post-treatment to collect information on safety (e.g., adverse events).
* Follow-up phase: From Day 29 post-treatment to Week 52 to collect information on VOD/SOS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory CD22-positive ALL
2. Patients who have never used BESPONSA before
3. Patients aged <18 years at the start of treatment with BESPONSA

Exclusion Criteria:

* None

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with relapsed or refractory CD22-positive ALL receiving BESPONSA
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-06-22 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | Up to 28 days after the last administration
Risk factors related to the onset of venoocclusive liver disease/sinusoidal obstruction syndrome | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1931035